CLINICAL TRIAL: NCT04913233
Title: Research on New Technologies for Screening and Early Diagnosis of Malignant Tumors - Establishment and Clinical Validation of New Technologies for Accurate Screening of Colorectal Cancer Based on Multi-omics
Brief Title: Establishment and Clinical Validation of New Technologies for Accurate Screening of Colorectal Cancer Based on Multi-omics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0199
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Cancer Screening; Colonoscopy; APCS; HRFQ
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

The current screening techniques for colorectal cancer include colonoscopy, fecal occult blood, and high-risk factor questionnaires. However, the colorectal cancer screening technology that has been widely used at present cannot take into account sensitivity and specificity, and the tumor detection rate is low.

The purpose of research:

1. Build a new type of population colorectal cancer precision screening technology program;
2. Improve the detection rate of colorectal cancer in the population by new methods (compared with the existing domestic advanced technology) by ≥20%, and improve the specificity of colorectal cancer screening by ≥15% without significantly reducing the sensitivity.

ELIGIBILITY:
Inclusion Criteria:

Age: 40-74 years old

Exclusion Criteria:

1. Combine severe disorders to make it unsuitable for colonoscopy
2. Combine other tumors
3. Mental and behavioral abnormalities do not cooperate with the screener
4. Researchers believe that other reasons are not suitable for enrollment

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals of 40-74 years old in non-high incidence of colorectal cancer areas(hospital outpatient population, community population in non-high-risk areas) .
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer detection rate in the population | through study completion, an average of 3 years
  Colorectal cancer detection rate in the population
Colorectal cancer screening specificity | through study completion, an average of 3 years
  Colorectal cancer screening specificity
Colorectal cancer screening sensitivity | through study completion, an average of 3 years
  Colorectal cancer screening sensitivity

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese Medicine Hospital of Haining City, Haining Cancer Preventional and Treatment Research Institute, Haining, Zhejiang
  - Jiashan County Cancer Prevention and Treatment Institute, Jiashan, Zhejiang
  - Lanxi City People's Hospital, Linjiang Hospital, Lanxi, Zhejiang